CLINICAL TRIAL: NCT04589559
Title: The Care After Life-threatening Medical Events (CALME) Pilot Study: An Investigation of Heart Rate Variability Biofeedback Training
Brief Title: The Care After Life-threatening Medical Events Study
Acronym: CALME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jeffrey Birk, Instructor in Medical Sciences, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS9001; P30AG064198 (NIH)
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Results first posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-07

CONDITIONS: Cardiac Arrest; Fear
Keywords: Cardiac arrest; Fear; Psychological distress; Heart Rate Variability Biofeedback
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: The intervention involves heart rate variability biofeedback (HRVB) administered via a smartphone app (Elite HRV) that receives real-time cardiac information from a chest-worn heart rate monitor (Polar H10).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: Heart Rate Variability Biofeedback (Experimental): Participants in this intervention group complete at-home heart rate variability biofeedback (HRVB) training using a chest-worn heart rate monitor and a smartphone app. They complete at least 10 minutes per day of HRVB training on at least 5 days per week for 3 weeks.
  Interventions: Behavioral: Heart Rate Variability Biofeedback Training

INTERVENTIONS:
Behavioral: Heart Rate Variability Biofeedback Training — First, participants are taught how to do relaxed, abdominal breathing. Second, they are taught how to breathe at a slow rate of 0.1 Hz (i.e., one completed breath cycle every 10 seconds). Third, they are taught how to monitor their heart rate variability (HRV) in real time using the smartphone app, which receives data wirelessly via Bluetooth from the heart rate monitor. Participants are instructed that their goal is to increase their HRV during the three weeks of at-home practice.
  Other Names: HRV Biofeedback

SUMMARY:
This study tests the feasibility of a home-based heart rate variability biofeedback (HRVB) intervention in survivors of cardiac arrest (CA). Specifically, the primary purpose of this pilot study is to assess feasibility, acceptability, appropriateness, usability, and compliance for an at-home, 3-week HRVB intervention in 10 participants. The study also tests whether cardiac-related interoceptive fear, trait anxiety, and negative affect decrease among CA survivors completing the HRVB intervention.

DETAILED DESCRIPTION:
HRV biofeedback is a technique that combines slow paced breathing with the use of accurate, moment-to-moment physiological monitoring. The goal is to make internal cardiac information available to people in order to help them learn how to increase the beat-to-beat variability in their heart's activity and thereby increase parasympathetic activity of the autonomic nervous system. Apart from active interventions such as exercise training that reliably increase HRV but that may be inappropriate for many cardiac patients, HRV biofeedback is an easy-to-implement technique which allows people to monitor and then ultimately alter their parasympathetic activity.

Research is needed to determine whether HRV biofeedback training has beneficial consequences for mental and cardiovascular health in patients who have experienced serious, life-threatening cardiac events. The investigator believes that cardiac arrest survivors, in particular, may stand to benefit from such an intervention because many of them experience clinically significant psychological distress after their medical event.

Distressed cardiac patients may be especially motivated to learn to influence their own heart activity in order to improve their own HRV, reduce their cardiovascular risk, and lessen their symptoms of psychological distress. Therefore, it may be wise to harness this motivation in the service of helping these patients deliberately learn to alter their own autonomic activity rather than simply breathing at a rate that automatically improves HRV without any learning process. By providing patients with an external (e.g., visual) form of feedback about their otherwise largely inaccessible autonomic physiology (i.e., vagus nerve activity), the investigator will conduct a feasibility study of HRV biofeedback training with the goal of increasing HRV and reducing anxiety symptoms.

The purpose of this pilot study is to examine the feasibility of enrolling 10 participants and assessing the feasibility, acceptability, appropriateness, and usability of the at-home, multi-week HRV biofeedback training as well as participants' compliance with the intervention. Additionally, the purpose of the study is to assess whether participants generally show a decrease in cardiac-related interoceptive fear, a decrease in trait anxiety, a decrease in negative affect, and an increase in HRV during the course of the study. The data collected from participants as part of this feasibility pilot will influence the decision to continue with a larger randomized clinical trial using the methods in this pilot together with a control group. Progress will be monitored with Polar H10 heart rate monitor - a supremely precise heart rate sensor that comes with the Polar Pro chest strap. It will be used with a smartphone app Elite HRV - which is non-experimental.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Fluent in English
3. A diagnosis of cardiac arrest (CA)
4. Time elapsed since their CA is less than 72 months
5. Elevated post-traumatic stress disorder (PTSD) symptom total scores on the 17-item Post-Traumatic Stress Disorder Checklist (PCL) of 30 or higher (i.e., greater than the median in a prior sample of cardiac arrest survivors) or elevated PCL-5 scores of 30 or higher or Acute Stress Disorder Scale (ASDS) scores of 34 or higher
6. Owns either an iPhone or Android smartphone in order to run the app involved in the intervention

Exclusion Criteria:

1. Breathing difficulty that does not allow participant to complete the intervention
2. Inability to comply with the protocol (either self-selected or indicated during screening that s/he could not complete all requested tasks). This includes, but is not limited to, patients with a level of cognitive impairment indicative of dementia and patients with current alcohol or substance abuse, and patients with severe mental illness (e.g., schizophrenia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Birk, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ten participants consented to participate in the study. All participants were assigned to the intervention condition in this single-arm feasibility study.
Groups:
- Intervention: Heart Rate Variability Biofeedback: Participants in this intervention group completed at-home heart rate variability biofeedback (HRVB) training using a wrist-worn heart rate monitor and a smartphone app. They were asked to complete at least 10 minutes per day of HRVB training on at least 5 days per week for 3 weeks.
  Heart Rate Variability Biofeedback Training: First, participants were taught how to do relaxed, abdominal breathing. Second, they were taught how to breathe at a slow rate of 0.1 Hz (i.e., one completed breath cycle every 10 seconds). Third, they were taught how to monitor their heart rate variability (HRV) in real time using the smartphone app, which received data wirelessly via Bluetooth from the heart rate monitor. Participants were instructed that their goal was to increase their HRV during the three weeks of at-home practice.
Period: Overall Study
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Heart Rate Variability Biofeedback: Participants in this intervention group complete at-home heart rate variability biofeedback (HRVB) training using a wrist-worn heart rate monitor and a smartphone app. They complete at least 10 minutes per day of HRVB training on at least 5 days per week for 3 weeks.
  Heart Rate Variability Biofeedback Training: First, participants are taught how to do relaxed, abdominal breathing. Second, they are taught how to breathe at a slow rate of 0.1 Hz (i.e., one completed breath cycle every 10 seconds). Third, they are taught how to monitor their heart rate variability (HRV) in real time using the smartphone app, which receives data wirelessly via Bluetooth from the heart rate monitor. Participants are instructed that their goal is to increase their HRV during the three weeks of at-home practice.
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.20 (15.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2
Sexual Orientation [Count of Participants; unit: Participants]
  Straight or heterosexual | 10
  Lesbian | 0
  Gay | 0
  Bisexual | 0
  Something else | 0
  Don't know / Not sure | 0
  Prefer not to say | 0
Partner Status [Count of Participants; unit: Participants]
  Single | 1
  Partner / Spouse | 6
  Separated | 1
  Widowed | 0
  Divorced | 2
  Prefer not to say | 0
Education [Count of Participants; unit: Participants]
  Less than high school | 0
  Some high school | 0
  High school diploma/GED | 0
  Trade school/Vocational school | 0
  Some college | 2
  College graduate | 3
  Graduate school/professional school | 5
  Prefer not to say | 0
Implanted Cardiac Device Type [Count of Participants; unit: Participants] — We assessed whether participants had an implanted cardiac device. Whereas pacemakers directly influence heart rate and heart rate variability, unpaced implantable cardioverter defibrillators generally do not, and unpaced cardiac monitors do not.
  Participants
    No cardiac device | 2
    Unpaced cardiac monitor | 1
    Implantable cardioverter defibrillator (ICD) | 4
    Pacemaker | 2
    Left ventricular assist device (LVAD) | 0
    Unknown or Not Reported | 1
Beta Blocker or Antiarrhythmic Medication [Count of Participants; unit: Participants] — We assessed whether participants were currently taking any beta-blocker medications or any antiarrhythmic medications. These medications are used to manage heart rhythm or to control blood pressure, among other uses.
  Participants
    Beta-Blockers | 6
    Antiarrhythmics | 0
    Neither Beta-Blockers nor Antiarrhythmics | 1
    Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Cardiac Arrest (CA) Survivors Whom we Approach Who Ultimately Agree to Participate in the Pilot Study
Description: This is to assess the feasibility of enrollment in the trial. The denominator for this metric is the number of potential participants who were approached and contacted by the study team who were determined to be eligible for the study. The numerator is the number of participants who enrolled in the study (i.e., 10 participants).
Time Frame: Baseline/Visit 1
Population: The population studied for this metric was the set of all potential participants who were approached and contacted by the study team and determined to meet the eligibility criteria for the study.
Measure: Number; unit: percentage of participants who enrolled
Groups:
- Intervention: Heart Rate Variability Biofeedback: Participants in this intervention group completed at-home heart rate variability biofeedback (HRVB) training using a chest-worn heart rate monitor and a smartphone app. They were asked to complete at least 10 minutes per day of HRVB training on at least 5 days per week for 3 weeks.
  Heart Rate Variability Biofeedback Training: First, participants were taught how to do relaxed, abdominal breathing. Second, they were taught how to breathe at a slow rate of 0.1 Hz (i.e., one completed breath cycle every 10 seconds). Third, they were taught how to monitor their heart rate variability (HRV) in real time using the smartphone app, which received data wirelessly via Bluetooth from the heart rate monitor. Participants were instructed that their goal was to increase their HRV during the three weeks of at-home practice.
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 12
percentage of participants who enrolled | 83.33

2. Secondary Outcome: Percentage of Enrolled Participants Who Complete the Pilot Study
Description: This is to assess successful program adherence.
Time Frame: Pre-training/Visit 2, Post-training/Visit 3 (approximately 3 weeks apart)
Measure: Number; unit: percentage of enrolled participants
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
percentage of enrolled participants | 100.0

3. Secondary Outcome: Percentage of Participants Who Complete a Majority of the At-home HRVB Sessions for the Pilot Study
Description: As a measure of intervention compliance, this is to assess the percentage of participants who complete a majority (>= 8 of 15) of the at-home HRVB sessions.
Time Frame: Pre-training/Visit 2, Post-training/Visit 3 (approximately 3 weeks apart)
Measure: Number; unit: percentage of enrolled participants
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
percentage of enrolled participants | 60.00

4. Secondary Outcome: Percentage of Participants Who Report Adequate Feasibility
Description: This is to assess the intervention's feasibility. The percentage of participants who report scores >= 4 for the feasibility total score reflects the percentage of participants who indicated that the intervention is adequately feasible.
Time Frame: Post-training/Visit 3 (approximately 3 weeks)
Measure: Number; unit: percentage of enrolled participants
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
percentage of enrolled participants | 90.00

5. Secondary Outcome: Percentage of Participants Who Report Adequate Acceptability
Description: This is to assess the intervention's acceptability. The percentage of participants who report scores >= 4 for the acceptability total score reflects the percentage of participants who indicated that the intervention is adequately acceptable.
Time Frame: Post-training/Visit 3 (approximately 3 weeks)
Measure: Number; unit: percentage of enrolled participants
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
percentage of enrolled participants | 90.00

6. Secondary Outcome: Percentage of Participants Who Report Adequate Appropriateness
Description: This is to assess the intervention's appropriateness for reducing anxiety, the proportion of participants who report scores >= 4 would be adequate.
  This is to assess the intervention's appropriateness for reducing anxiety. The percentage of participants who report scores >= 4 for the appropriateness-for-reducing-anxiety total score reflects the percentage of participants who indicated that the intervention is adequately appropriate for reducing anxiety.
Time Frame: Post-training/Visit 3 (approximately 3 weeks)
Measure: Number; unit: percentage of enrolled participants
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
percentage of enrolled participants | 80.00

7. Secondary Outcome: Percentage of Participants Who Report Adequate Usability
Description: We will assess the percentage of participants who report total scores >= 68 for their rating of the intervention's usability using the System Usability Scale.
Time Frame: Post-training/Visit 3 (approximately 3 weeks)
Measure: Number; unit: percentage of enrolled participants
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
percentage of enrolled participants | 80.00

8. Secondary Outcome: Visit-2-to-3 Change in Cardiac-related Interoceptive Fear
Description: This is to assess the Visit-2-to-3 change in cardiac-related interoceptive fear measured as the within-person difference in the sum of the four cardiac-related items from the physical subscale of the Anxiety Sensitivity Index. The total score ranges from a minimum of 0 units on a scale to a maximum of 16 units on a scale. Lower scores indicate lower anxiety.
Time Frame: Pre-training/Visit 2, Post-training/Visit 3 (approximately 3 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
score on a scale | -1.50 (3.03)
Statistical Analysis 1: Comparison: Intervention: Heart Rate Variability Biofeedback; Test type: Other — Paired-samples t-test; p = 0.152, t-test, 2 sided; Paired-samples t-test; Mean change score = -1.50, 95% CI 2-sided [-3.67 to 0.67] — A negative value of the estimation parameter of mean change score indicates a reduction in cardiac-related interoceptive fear

9. Secondary Outcome: Visit-2-to-3 Change in Trait Anxiety
Description: This is to assess the Visit-2-to-3 change in trait anxiety measured as the within-person difference in the total score of the trait version of the State-Trait Anxiety Inventory. The total score ranges from a minimum of 20 units on a scale to a maximum of 80 units on a scale. Higher scores indicate higher anxiety.
Time Frame: Pre-training/Visit 2, Post-training/Visit 3 (approximately 3 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
score on a scale | -6.20 (7.70)
Statistical Analysis 1: Comparison: Intervention: Heart Rate Variability Biofeedback; Test type: Other — Paired-samples t-test; p = 0.031, t-test, 2 sided; Paired-samples t-test; Mean change score = -6.20, 95% CI 2-sided [-11.71 to -0.69] — A negative value of the estimation parameter of mean change score indicates a reduction in trait anxiety

10. Secondary Outcome: Visit-2-to-3 Change in Trait Negative Affect
Description: This is to assess the Visit-2-to-3 change in trait negative affect measured as the within-person difference in the total score of the negative subscale of the Positive and Negative Affect Schedule. The total score ranges from a minimum of 10 units on a scale to a maximum of 50 units on a scale. Lower scores represent lower levels of Negative Affect.
Time Frame: Pre-training/Visit 2, Post-training/Visit 3 (approximately 3 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
score on a scale | -1.90 (5.74)
Statistical Analysis 1: Comparison: Intervention: Heart Rate Variability Biofeedback; Test type: Other — Paired-samples t-test; p = 0.323, t-test, 2 sided; Paired-samples t-test; Mean change score = -1.90, 95% CI 2-sided [-6.01 to 2.21] — A negative value of the estimation parameter of mean change score indicates a reduction in negative affect

11. Secondary Outcome: Heart Rate Variability (HRV)
Description: This is to assess HRV using participants' exported and deidentified data from the Elite HRV smartphone app. Specifically, HRV is operationalized as the natural log of the root mean square of the successive difference (lnRMSSD), a standard measure of beat-to-beat HRV. This HRV measure is recorded for each at-home training session completed by participants using the app and the heart rate monitor.
Time Frame: Up to 3 weeks (starting after Visit 2 and extending until Visit 3)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Intervention: Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
milliseconds | 0.58 (1.04)
Statistical Analysis 1: Comparison: Intervention: Heart Rate Variability Biofeedback; Test type: Other — Paired-samples t-test; p = 0.112, t-test, 2 sided; Paired-samples t-test; Mean change in the measure = 0.58, 95% CI 2-sided [-0.16 to 1.33] — A positive value of the estimation parameter of mean change in the measure indicates an increase in heart rate variability

ADVERSE EVENTS:
Time Frame: Adverse events were assessed over the full study assessment period that lasted approximately 4 weeks total, from Visit 1 to Visit 3 of the study.
Arm/Group | Intervention: Heart Rate Variability Biofeedback
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT04589559/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT04589559/SAP_001.pdf